CLINICAL TRIAL: NCT03847727
Title: Study of Bendamustine and Rituximab as Induction Immunochemotherapy Followed by Maintenance Bendamustine and Rituximab in Relapsed and Refractory B-cell Chronic Lymphocytic Leukemia (CLL)
Brief Title: Bendamustine and Rituximab (BR) as Induction and Maintenance in Relapsed and Refractory Chronic Lymphocytic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: RSMU-CLL-2013
Record Dates: First submitted 2019-01-15; First posted 2019-02-20 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Bendamustine Hydrochloride; Rituximab; Maintenance
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Maintenance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: 6 cycles BR -> 4 x BR: Induction plus BR as maintenance (N=56)
  Interventions: Drug: BR as Maintenance
- Proper historical control: 6 cycles BR: Induction only (N=56)

INTERVENTIONS:
Drug: BR as Maintenance — Patients of the study group who have achieved at least a partial response after 6 cycles of BR induction will receive additionally 4 cycles of BR every 3 months as maintenance therapy.
  Groups: Experimental: 6 cycles BR -> 4 x BR

SUMMARY:
CLL is an incurable disease with conventional chemotherapy. In the absence of TP53 disruption, a chemoimmunotherapy (CIT) regimen is recommended as front-line and second-line treatment in those patients who attained a long progression-free survival (PFS) with the previous regimen. Bendamustine and rituximab (BR) is one of the most widely adopted CIT regimens, including second-line treatment. Unfortunately, durations of remission following BR combination therapy tend to be short in patients with heavily pre-treated disease or who have already received rituximab. The incorporation of a maintenance following induction chemotherapy to overcome the shorter remission durations in this population is a reasonable option.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CD20-positive CLL that meets the iwCLL criteria (Hallek et al, 2008).
* Relapsed or refractory status of disease after at least one prior chemotherapy regimen.
* ECOG performance status of 0-2 at study entry
* Patients have not received prior therapy with bendamustine
* Prior therapy with rituximab is permitted, even in the setting of rituximab refractory disease.

For inclusion in the research part of maintenance therapy (phase B):

* At least a partial response (PR or better; Hallek et al, 2008) must be achieved after induction of BR (phase A)

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent document or complying with the protocol treatment.
* Pregnant or breast-feeding females.
* Known to be positive for human immunodeficiency virus (HIV) or infectious hepatitis (type B or C).
* Patients are not eligible if there is a prior history or current evidence of central nervous system or leptomeningeal involvement.
* Richter syndrome or chronic prolymphocytic leukemia.
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia.
* Concurrent use of other anti-cancer agents or treatments.
* Laboratory test results within these ranges: ANC ≤ 1000/μL, Platelet count ≤ 75,000/μL.
* Total bilirubin Total bilirubin ≥ 2X upper limit laboratory normal (ULN). Patients with non-clinically significant elevations of bilirubin due to Gilbert's disease are not required to meet these criteria.
* Serum transaminases AST (SGOT) and ALT (SGPT) ≥ 3 x ULN, and/or serum alkaline phosphatase ≥ 5 X ULN.
* New York Heart Association class 3-4 heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed or refractory CLL receiving treatment at the University Hematology Hospital and Ambulant clinic.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2020-12-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 42 months
  PFS is defined as the number of days from the date of first dose of any study drug (rituximab or bendamustine) to the date of disease progression or death, whichever occurs first. PFS will be compared with its proper historical control (BR as induction without subsequent maintenance).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Approximately 24 months after initial dose of study drug.
  ORR is defined as the proportion of participants with an overall response (CR, CRi, nodular partial remission [nPR] plus partial remission [PR]) per the 2008 Modified IWCLL NCI-WG criteria.
Overall Survival (OS) | 60 months (6 months induction therapy, 12 months maintenance, 42 months long-term follow-up
  OS is defined as number of days from the date of first dose of any study drug (rituximab or bendamustine) to the date of death.
Safety evaluations | Up to 30 months
  To determine the safety and tolerability of induction chemotherapy and maintenance therapy separately for two groups as assessed by CTCAE v4.0:
Health Related Quality of Life (HRQoL) | Up to 30 months
  To determinate the effect of maintenance therapy on HRQoL using the EORTC Core quality of life questionnaire (QOL-C30, version 3.0).

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Semochkin, Professor, Principal Investigator — Pirogov Russian National Research Medical University
Locations (1):
- Semochkin Sergey, Moscow, Ostrovitianov Str. 1, Russia